CLINICAL TRIAL: NCT02303223
Title: Propofol Pharmacokinetics in Children After Single Bolus Dose
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Naveen Naik, Post graduate resident, Post Graduate Institute of Medical Education and Research, Chandigarh
Organization: PIMERIndia (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: NK/MD/1008/13592-93
Record Dates: First submitted 2014-10-26; First posted 2014-11-27 (Estimated); Last update posted 2015-01-30 (Estimated); Status verified 2015-01

CONDITIONS: Propofol Pharmacokinetics
MeSH Terms: interventions — Propofol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Propofol (Other): Single intravenous bolus dose of Propofol 2.5mg/kg for induction of anesthesia
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Propofol

SUMMARY:
The principle objective of this study is to evaluate pharmacokinetics of propofol after single iv bolus dose in 12 Indian children and to develop a simple pharmacokinetic model of propofol.

DETAILED DESCRIPTION:
PROPOFOL is the most suitable agent currently available for induction and maintenance of anesthesia. So far, the pharmacokinetics of propofol has not been studied in Indian children. We believe that this pharmacokinetic characterization of propofol will help in better management of these patients undergoing surgery under total intravenous anesthesia (TIVA) in our setup. 12 ASA (American Society of Anesthesiologists) grade I patients, 5 to 12 years old planned for elective surgery will be included. Premedication will be done with syrup midazolam 0.5mg/kg. After shifting the patient to the operation table, routine physiological monitoring will be commenced and two intravenous lines will be secured,one in the antecubital vein of one arm and the other vein on the dorsum of the contralateral hand. The antecubital venous access will be used for blood sampling. Anesthetic technique will consist of fentanyl bolus dose of 2ug/kg followed by propofol bolus dose of 2.5 mg/kg. No further propofol will be administered. After loss of consciousness , patients will be paralysed with atracurium (0.5mg/kg) and endotracheal intubation will be performed. Anesthesia will be maintained with isoflurane, oxygen (50%) and nitrous oxide (50%), and intermittent dosages of atracurium. A total of twelve samples will be collected from each patient at 0, 2, 4, 6, 10, 20, 30, 60, 90, 120, 240, and 480 min after administration of bolus dose of propofol.The samples will be analyzed using a modified High Performance Liquid Chromatography method described by Pavan et al. The pharmacokinetic parameters will be evaluated using three compartment model to develop a pharmacokinetic model by using the software WINNONLIN (Windows Non Linear Regression Program).

ELIGIBILITY:
Inclusion Criteria:

* Children aged 5-12 years and ASA (American Society of Anesthesiologists) grade I, planned for elective surgery under general anesthesia

Exclusion Criteria:entered

* Allergic history to one of the constituents of propofol
* Any evidence of cardiovascular, respiratory,metabolic ,renal ,hematologic,hepatic or central nervous system disease
* Previous adverse anesthetic events
* Potential airway management problems

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2014-01; Primary Completion 2014-12 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Plasma Propofol concentration | 0, 2, 4, 6, 10, 20, 30, 60, 90, 120, 240 and 480 minutes post loading dose of Propofol

CONTACTS AND LOCATIONS:
Overall Officials: Goverdhan D Puri, MD, Study Director — Post Graduate Institute of Medical Education and Research, Chandigarh
Locations (1):
- Post Graduate Institute of Medical Education and Research, Chandigarh, Chandigarh, India

REFERENCES:
- [Background] Kataria BK, Ved SA, Nicodemus HF, Hoy GR, Lea D, Dubois MY, Mandema JW, Shafer SL. The pharmacokinetics of propofol in children using three different data analysis approaches. Anesthesiology. 1994 Jan;80(1):104-22. doi: 10.1097/00000542-199401000-00018. PMID 8291699
- [Background] Pavan I, Buglione E, Massiccio M, Gregoretti C, Burbi L, Berardino M. Monitoring propofol serum levels by rapid and sensitive reversed-phase high-performance liquid chromatography during prolonged sedation in ICU patients. J Chromatogr Sci. 1992 May;30(5):164-6. doi: 10.1093/chromsci/30.5.164. PMID 1322421
- [Background] Marsh B, White M, Morton N, Kenny GN. Pharmacokinetic model driven infusion of propofol in children. Br J Anaesth. 1991 Jul;67(1):41-8. doi: 10.1093/bja/67.1.41. PMID 1859758